CLINICAL TRIAL: NCT05361187
Title: STRAIT: Evaluation of Safety and Performance of the BOBBY™ Balloon Guide Catheter for Endovascular Treatment of Acute Ischemic Stroke
Brief Title: BOBBY™ Balloon Guide Catheter for Endovascular Treatment of Acute Ischemic Stroke
Acronym: STRAIT
Status: Terminated | Type: Observational
Why Stopped: endpoint reached
Sponsor: Microvention-Terumo, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: STRAIT
Record Dates: First submitted 2022-04-13; First posted 2022-05-04 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Cerebrovascular Stroke
Keywords: Cerebrovascular Stroke; Thrombectomy; Balloon Guide Catheter
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- single arm, observational post market study: Patients with an acute ischemic stroke with treatment including the BOBBY™ BGC
  Interventions: Device: BOBBY™ Balloon Guide Catheter intended for use in neurovascular procedures, performing or as an adjunctive device

INTERVENTIONS:
Device: BOBBY™ Balloon Guide Catheter intended for use in neurovascular procedures, performing or as an adjunctive device — The BOBBY™ BGC used during a mechanical thrombectomy procedure (stent retriever alone, contact aspiration alone or stent retriever and contact aspiration) and according to the instruction for use (IFU).

SUMMARY:
Evaluation of the safety and performance of the BOBBY™ Balloon Guide Catheter (BGC) in patients with an acute ischemic stroke treatment, a sudden reduction or termination of the blood circulation of the brain, caused by a clot. Immediate treatment is needed to restore the blood circulation in the brain, performing a mechanical removal of the clot (thrombectomy). To prevent clot particles migrating in other parts of the brain circulation during the thrombectomy, balloon guiding catheters are inserted. The aim of the study is to evaluate the safety and performance of the balloon guide catheter BOBBY™ by collecting information from patients, treated with a mechanical thrombectomy and the balloon guide catheter (BOBBY™) after acute ischemic stroke

DETAILED DESCRIPTION:
The main objective of the STRAIT study is to assess the performance of the mechanical thrombectomy using a BOBBY™ Balloon Guide Catheter (BGC) as adjunctive device for endovascular treatment of patients suffering from an anterior circulation acute ischemic stroke. Interventional procedures and clinical follow-up will be performed per standard of care. Patient health-related and imaging data will be collected as of stroke onset time up to 90 days follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 and ≤ 85 years of age
* Informed consent by the patient or legal authorized representative for data collection is obtained
* Patient eligible for the mechanical thrombectomy treatment with adjunctive use of the BOBBY™ BGC
* Patient presenting with an anterior circulation large-vessel occlusion of distal internal carotic artery (ICA ) through proximal M2 confirmed by computed tomograph angiography (CTA), magnetic resonance angiography (MRA), or digital subtraction angiography (DSA).
* Core-infarct volume of Alberta Stroke Program Early CT Score (ASPECTS) ≥ 6 based on baseline CT or MR imaging
* Treatment initiated (groin puncture) within 8 hours of symptom onset.
* Patient with a pre-treatment National Institutes of Health Stroke Scale (NIHSS) score ≥5
* Patient with no personal condition disabling the site to contact him/her at 90 days after procedure

Exclusion Criteria:

* Patient has evidence of cerebral ischemia in the posterior circulation
* Patient presents severe unilateral or bilateral carotid artery stenosis requiring stent treatment during the procedure
* Pregnancy or breastfeeding
* Patient presents other serious medical illness (e.g., cancer) with estimated life expectancy of less than 3 months
* Patient has a planned procedure that may cause non-compliance with the protocol or confound data interpretation
* Patient is already participating in an investigational drug or device trial (change routine care of the patient)
* Patient has evidence of intracerebral hemorrhage on initial imaging
* Patient has a significant mass effect with midline shift

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from an anterior circulation acute ischemic stroke eligible to mechanical thrombectomy using a BOBBY™ Balloon Guide Catheter will be screened consecutively by the enrolling center. The patients will be selected in accordance with inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the proportion of patients with successful reperfusion defined as mTICI≥2b per Core Laboratory evaluation. | 90 days
  Successful reperfusion defined as mTICI≥2b by independent Core Laboratory evaluation.

SECONDARY OUTCOMES:
Technical success: successful placement of the BOBBY™ BGC at the skull base | 90 days
  Bobby catheter placement evaluated at predefined segments (cervical, petrous, cavernous, paraclinoid) of the internal carotic artery (ICA) per independent Core Laboratory evaluation
Near complete reperfusion defined as mTICI≥2c | 90 days
  mTICI evaluation per independent Core Lab members
Patients with modified First Pass Effect observed (mFPE: mTICI≥2b after one pass) | 90 days
  mTICI result after first pass evaluated by independent Core Lab members
90 days post-procedure modified Ranking Scale (mRS) | 90 days
  modified Ranking Scale (mRS) assessment and questionnaire at 90 days follow up visit.
  The mRS has a scale from 0 till 6. 0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead
Mortality at 24 hours and 90 days | 24 hours and 90 days
  Serious adverse event evaluation validated by clinical event committee
Safety evaluation device malfunction | 90 days
  Device related adverse event evaluation and follow up, validated by clinical event committee
NIHSS at 24h post-procedure | 24 hours
  NIHSS (National Institut Health Stroke Scale) evaluation by questionnaire to assess worsening of condition compared to baseline.
  The NIHSS score covers 11 specific ability items. Each item can been scored between 0 and 4, with 0 indicating a normal function and higher scores indicating the lever of impairment. The total summ of all the ablity items is the total NIHSS score. The maximum possible score is 42, with the minimum score being a 0.
  0 No stroke symptoms, 1-4, Minor stroke, 5-15 Moderate stroke,16-20 Moderate to severe stroke, 21-42 Severe stroke
Procedure related events | 24 hours
  Procedure related events and outcome evaluation validated
Occurence of new territory embolization | 24 hours
  Assessment by independent Core Lab members of DSA or MRA at the end of the procedure and at 24 hours
Occurrence of symptomatic intracranial hemorrhage (sICH) within 24 hours | 24 hours
  procedure imaging assessment of imaging

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Boeckh-Behrens, MD, Principal Investigator — Neuro-Kopf-Zentrum Klinikum rechts der Isar der Technischen Universität; Patricia Boyer, Study Director — Microvention-Terumo, Inc.
Locations (9):
- Germany (6):
  - Neuro-Kopf-Zentrum Klinikum rechts der Isar der Technischen Universität München, Munich, Bavaria
  - Martin Luther Universität Halle, Halle, Halle
  - Neurologische Klinik Abteilung für Neuroradiologie, Heidelberg
  - Klinikum Ingolstadt, Zentrum für Radiologie und Neuroradiologie, Ingolstadt
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - Department of Neuroradiology, University Hospital of Paracelsus Medical Private University, Nuremberg
- Switzerland (3):
  - Devision Neuroradiology, Kantonsspital Aarau, Aarau
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne
  - Department of Neuroradiology, University hospital Zürich, Zurich